CLINICAL TRIAL: NCT06314204
Title: Impact of Cannabis Consumption on the Course, Modalities of Hospitalization and the Short-term Prognosis of Inpatients Suffering From Psychotic Symptoms : Multicenter Comparative Observational Study
Brief Title: Impact of Cannabis Consumption on the Course, Modalities of Hospitalization and the Short-term Prognosis of Inpatients Suffering From Psychotic Symptoms
Acronym: canhope
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Noomane Bouaziz, MD, MBBS, psychiatrist and investigator, Centre hospitalier de Ville-Evrard, France
Other Study IDs: 2015-A01222-47
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Psychotic; Disorder, Cannabis
Keywords: cannabis-Timing-hospitalization-psychotic sympyomatology
MeSH Terms: conditions — Mental Disorders; Marijuana Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Few studies have evaluated, in patients with symptomatology the impact of cannabis use on the duration of hospitalization and on short- and medium-term developments. The objective of this study will be to assess the impact of cannabis on the duration, the hospitalization and the short- and medium-term evolution of patients with psychotic symptoms and cannabis use. We hypothesize that these patients (in comparison with patients with psychotic symptomatology and not using cannabis) would be hospitalized more long, exposed to a higher risk of resistance to the usual therapeutics, would have a lack of therapeutic alliance and insight, relapses and hospitalizations more frequent, more marked negative symptoms and lower quality remission. They would also be more prone to impulsive and aggressive behaviour.

DETAILED DESCRIPTION:
Several studies have reported that cannabis use worsen the prognosis of psychiatric pathologies in general and psychotic in particular.

Few or no studies have evaluated the impact of cannabis consumption on patients with psychotic symptoms during their hospitalization (duration, type of hospitalization, quality of relationship with staff hospital), and on the short-term prognosis.

The objective of this study will be to assess the impact of cannabis on the duration of the hospitalization and the short- and medium-term evolution of patients with a psychotic symptomatology and cannabis use. Making the hypothesis that these patients (compared to patients with symptomatology psychotic and not using cannabis) would be hospitalized longer, exposed at a higher risk of resistance to the usual therapies, to have a lack of alliance therapeutic and insight, relapses and more frequent hospitalizations and symptoms.

They would also be more likely to have lower quality. They would also be more likely to be impulsive, and have aggressive behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in psychiatry regardless of the mode of hospitalization
* With or without protective measures (guardianship or curatorship)
* Presenting psychotic symptoms (schizophrenia, schizo affective disorder, thymic disorder with psychotic characteristic, psychotic disorder substance-induced, brief psychotic disorder, schizophrenic disorders, delirious disorders)
* Members of the social security system
* Enlightened information

Exclusion Criteria:

* Degenerative neurological pathologies or mental retardation
* Psychotic disorders secondary to generalized medical conditions(epilepsy, delirium tremens, tumors, etc.)
* Other psychiatric pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study will consist of patients over the age of 18 with trans-nosographic psychotic symptomatology (schizophrenia, schizoaffective disorder, mood disorder with psychotic characteristic, psychotic disorder induced by substances, brief psychotic disorder, schizophrenic disorder, delirious disorders), hospitalized in psychiatry, free care or under duress in the Hospitalization Units to Full-time (UHTP) EPS Ville-Evrard. This protocol also concerns protected adults. Forecasted number of patients: 200 patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09-20 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
PANSS: Positive and Negative Syndrom Scale | AT the beginning of the study, before any procedure, (T1)
  This scale permit to assess the severity of schizophrenia.Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112. The total PANSS score is simply the sum of the sub scales.
PANSS: Positive and Negative Syndrom Scale | Approximatively 2 or 3 weeks after T1,On the day of the discharge (T2)
  This scale permit to assess the severity of schizophrenia.Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112. The total PANSS score is simply the sum of the sub scales.
PANSS: Positive and Negative Syndrom Scale | 1 month after the discharge (T3)
  This scale permit to assess the severity of schizophrenia.Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112. The total PANSS score is simply the sum of the sub scales.
PANSS: Positive and Negative Syndrom Scale | 3 month after the discharge (T4)
  This scale permit to assess the severity of schizophrenia.Positive Scale, Negative Scale, and General Psychopathology Scale. Each subscale is rated with 1 to 7 points ranging from absent to extreme. The range for the Positive and Negative Scales is 7-49, and the range for the General Psychopathology Scale is 16-112. The total PANSS score is simply the sum of the sub scales.
MCQ-SF :Marijuana Craving Questionnaire- Short Form | AT the beginning of the study, before any procedure (T1)
  The scale permit to determine the marijuana craving. The subscales exhibited low to moderate, positive intercorrelations and were significantly correlated with marijuana use history and a wide range of single-item measures of craving. Conclusions. Findings suggested that four specific constructs characterize craving for marijuana: (1) compulsivity, an inability to control marijuana use; (2) emotionality, use of marijuana in anticipation of relief from withdrawal or negative mood; (3) expectancy, anticipation of positive outcomes from smoking marijuana; and (4) purposefulness, intention and planning to use marijuana for positive outcomes.
MCQ-SF :Marijuana Craving Questionnaire- Short Form) | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  The scale permit to determine the marijuana craving. The subscales exhibited low to moderate, positive intercorrelations and were significantly correlated with marijuana use history and a wide range of single-item measures of craving. Conclusions. Findings suggested that four specific constructs characterize craving for marijuana: (1) compulsivity, an inability to control marijuana use; (2) emotionality, use of marijuana in anticipation of relief from withdrawal or negative mood; (3) expectancy, anticipation of positive outcomes from smoking marijuana; and (4) purposefulness, intention and planning to use marijuana for positive outcomes.
MCQ-SF :Marijuana Craving Questionnaire- Short Form) | one month after the discharge
  The scale permit to determine the marijuana craving. The subscales exhibited low to moderate, positive intercorrelations and were significantly correlated with marijuana use history and a wide range of single-item measures of craving. Conclusions. Findings suggested that four specific constructs characterize craving for marijuana: (1) compulsivity, an inability to control marijuana use; (2) emotionality, use of marijuana in anticipation of relief from withdrawal or negative mood; (3) expectancy, anticipation of positive outcomes from smoking marijuana; and (4) purposefulness, intention and planning to use marijuana for positive outcomes.
MCQ-SF :Marijuana Craving Questionnaire- Short Form) | three month after the discharge
  The scale permit to determine the marijuana craving. The subscales exhibited low to moderate, positive intercorrelations and were significantly correlated with marijuana use history and a wide range of single-item measures of craving. Conclusions. Findings suggested that four specific constructs characterize craving for marijuana: (1) compulsivity, an inability to control marijuana use; (2) emotionality, use of marijuana in anticipation of relief from withdrawal or negative mood; (3) expectancy, anticipation of positive outcomes from smoking marijuana; and (4) purposefulness, intention and planning to use marijuana for positive outcomes.
CGI: Clinical Global Impression | AT the beginning of the study, before any procedure (T1)
  It is used with all patients, allowing the evaluation of the improvement of assessing the severity and change of the overall clinical condition.
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  Improvement scale The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
CGI: Clinical Global Impression | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  It is used with all patients, allowing the evaluation of the improvement of assessing the severity and change of the overall clinical condition.
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  Improvement scale The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
CGI: Clinical Global Impression | one month after the discharge
  It is used with all patients, allowing the evaluation of the improvement of assessing the severity and change of the overall clinical condition.
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  Improvement scale The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
CGI: Clinical Global Impression | three month after the discharge
  It is used with all patients, allowing the evaluation of the improvement of assessing the severity and change of the overall clinical condition.
  The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  Improvement scale The clinical global impression - improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
MADRS: Montgomery Åsberg Depression Rating Scale | AT the beginning of the study, before any procedure (T1)
  It is validated in France by Pellet and its collaborators in 1987. It allows to evaluate the modifications of mood.
  It has 10 psychic and somatic items (apparent sadness, sadness expressed, inner tension, insomnia, loss of appetite, difficulty concentrating, weariness, loss of feelings, pessimism and thoughts of suicide) sides from 0 to 6 according to the 6 degrees of severity and whose scores add up.
MADRS: Montgomery Åsberg Depression Rating Scale | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  It is validated in France by Pellet and its collaborators in 1987. It allows to evaluate the modifications of mood.
  It has 10 psychic and somatic items (apparent sadness, sadness expressed, inner tension, insomnia, loss of appetite, difficulty concentrating, weariness, loss of feelings, pessimism and thoughts of suicide) sides from 0 to 6 according to the 6 degrees of severity and whose scores add up.
MADRS: Montgomery Åsberg Depression Rating Scale | one month after the discharge
  It is validated in France by Pellet and its collaborators in 1987. It allows to evaluate the modifications of mood.
  It has 10 psychic and somatic items (apparent sadness, sadness expressed, inner tension, insomnia, loss of appetite, difficulty concentrating, weariness, loss of feelings, pessimism and thoughts of suicide) sides from 0 to 6 according to the 6 degrees of severity and whose scores add up.
MADRS: Montgomery Åsberg Depression Rating Scale | Three month after the discharge
  It is validated in France by Pellet and its collaborators in 1987. It allows to evaluate the modifications of mood.
  It has 10 psychic and somatic items (apparent sadness, sadness expressed, inner tension, insomnia, loss of appetite, difficulty concentrating, weariness, loss of feelings, pessimism and thoughts of suicide) sides from 0 to 6 according to the 6 degrees of severity and whose scores add up.
PDS: Psychotic Depression Scale | AT the beginning of the study, before any procedure (T1)
  It is composed of 32 items. Among the PDS items, those related to the "mood" factors depressive" (8 items) and "vegetative signs" (3 items) allow an evaluation of the depression regardless of negative symptoms or extrapyramidal symptoms.
  All items are scoring from 0 to 6:
  0: nothing 2 :light 4: important 6: extreme
PDS: Psychotic Depression Scale | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  It is composed of 32 items. Among the PDS items, those related to the "mood" factors depressive" (8 items) and "vegetative signs" (3 items) allow an evaluation of the depression regardless of negative symptoms or extrapyramidal symptoms.
  All items are scoring from 0 to 6:
  0: nothing 2 :light 4: important 6: extreme
PDS: Psychotic Depression Scale | one month after the discharge
  It is composed of 32 items. Among the PDS items, those related to the "mood" factors depressive" (8 items) and "vegetative signs" (3 items) allow an evaluation of the depression regardless of negative symptoms or extrapyramidal symptoms. The overall PDS score is correlated to the overall MADRS scores.
  All items are scoring from 0 to 6:
  0: nothing 2 :light 4: important 6: extreme
PDS: Psychotic Depression Scale | Three month after the discharge
  It is composed of 32 items. Among the PDS items, those related to the "mood" factors depressive" (8 items) and "vegetative signs" (3 items) allow an evaluation of the depression regardless of negative symptoms or extrapyramidal symptoms. The overall PDS score is correlated to the overall MADRS scores.
  All items are scoring from 0 to 6:
  0: nothing 2 :light 4: important 6: extreme
YMRS: Young Mania Rating Scale | AT the beginning of the study, before any procedure (T1)
  The YMRS is a scale of 11 questions to assess the severity of symptoms maniacs. It is considered the gold standard of scales evaluating mania.
  This instrument is widely used both in the clinic and in research. It is appropriate both to assess the initial severity of manic symptoms, and the response to treatment in patients with bipolar disorder type I and II. Each item of YMRS given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
  There are well described anchor points for each grade of severity.
YMRS: Young Mania Rating Scale | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  The YMRS is a scale of 11 questions to assess the severity of symptoms maniacs. It is considered the gold standard of scales evaluating mania.
  This instrument is widely used both in the clinic and in research. It is appropriate both to assess the initial severity of manic symptoms, and the response to treatment in patients with bipolar disorder type I and II. Each item of YMRS given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
  There are well described anchor points for each grade of severity.
YMRS: Young Mania Rating Scale | one month after the discharge
  The YMRS is a scale of 11 questions to assess the severity of symptoms maniacs. It is considered the gold standard of scales evaluating mania.
  This instrument is widely used both in the clinic and in research. It is appropriate both to assess the initial severity of manic symptoms, and the response to treatment in patients with bipolar disorder type I and II. Each item of YMRS given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
  There are well described anchor points for each grade of severity.
YMRS: Young Mania Rating Scale | Three month after the discharge
  The YMRS is a scale of 11 questions to assess the severity of symptoms maniacs. It is considered the gold standard of scales evaluating mania.
  This instrument is widely used both in the clinic and in research. It is appropriate both to assess the initial severity of manic symptoms, and the response to treatment in patients with bipolar disorder type I and II. Each item of YMRS given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
  There are well described anchor points for each grade of severity.
CDS: Self-Consciousness Revised Scale | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  This scale represents a cross-cultural validation in of the Self-Consciousness Revised Scale by Scheier et al. This scale measures three aspects of the self-awareness, that is, private, public self-awareness and social anxiety. It includes 22 statements. The scale is rating 0-3 point:
  0: not at all like me
  1. a little bit like me
  2. quite similar to me
  3. Very much like me . The time to complete will be 10 minutes.
CTQ: Childhood Trauma Questionnaire | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  The Child Trauma Questionnaire is a questionnaire developed by Bernstein et al. (1994) which includes 70 items with a scale of type Likert in five answer choices (from 1 = "never true" to 5 = "very often true").
  It was developed from a detailed review of the literature on abuse and also from experience a structured interview, the Childhood Trauma Interview, developed by the same authors. The ten minutes will be required.
BFI: Big Five Inventory | Approximatively 2 or 3 weeks after T1 ,On the day of the discharge (T2)
  The Personality Dimension Scale, BIG FIVE, FFS: John et al. developed the Big Five Inventory (BFI). This consists of 44 items in its American version, consisting of short phrases based on the adjectives of traits known to be the prototype markers of the "Big Five" John et al. no longer denotes the factors but assigns them a letter accompanied by a set of explanatory and synthetic terms of the definition: E (Extraversion, Energy, Enthusiasm); A (Agreeability, Altruism, Affection); C (Consciousness, Control, Constraint); N (Negative Emotions, Neuroticism, Nervousness); O (Openness, Originality, Openness).
  The Time of passing is 10 minutes.
  1. disagree strongly
  2. disagree a little
  3. Neither agree or nor disagree
  4. agree a little
  5. agree strongly

CONTACTS AND LOCATIONS:
Locations (1):
- unité de recherche clinique de l'E.P.S de Ville Evrard, Neuilly-sur-Marne, France